CLINICAL TRIAL: NCT02636348
Title: Evaluation of Calcium and Vitamin D Supplementation for Optimizing Bone Health During Marine Corps Recruit Training
Brief Title: Evaluation of Calcium and Vitamin D Supplementation During Marine Corps Training
Acronym: MCRD-PI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15-21-HC
Record Dates: First submitted 2015-06-24; First posted 2015-12-21 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Nutrition Status; Bone Health
Keywords: Calcium; Vitamin D
MeSH Terms: interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Calcium/Vitamin D Bar (Experimental): Dietary supplement consumed as 2 calcium and vitamin D fortified snack bars per day
  Interventions: Dietary Supplement: Calcium/Vitamin D
- Calcium/Vitamin D Pill (Experimental): Dietary supplement consumed as several capsules per day
  Interventions: Dietary Supplement: Calcium/Vitamin D
- Placebo Bar (Placebo Comparator): Placebo consumed as 2 isocaloric, unfortified snack bars per day
  Interventions: Dietary Supplement: Placebo
- Placebo Pill (Placebo Comparator): Placebo consumed as several capsules per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Calcium/Vitamin D — 2000 mg calcium and 1000 IU vitamin D administered daily as 8 pills or 2 fortified snack bars.
  Arms: Calcium/Vitamin D Bar; Calcium/Vitamin D Pill
Dietary Supplement: Placebo — Administered daily as 8 placebo pills or 2 unfortified snack bars.
  Arms: Placebo Bar; Placebo Pill

SUMMARY:
The primary objective of this randomized, double-blind, placebo-controlled trial is to determine the efficacy and effectiveness of Ca and vitamin D supplementation provided daily throughout Marine Corps recruit training on maintenance of PTH and indices of bone strength in Marine Corps recruits. The investigators hypothesize that Ca+D will prevent elevations in PTH and result in greater increases in indices of bone strength compared to placebo.

DETAILED DESCRIPTION:
Military recruits undergoing initial military training (IMT) are 17 times more likely to develop stress fractures compared to active duty service members. Up to 800 male and female recruits will be enrolled at the MCRD, Parris Island, SC over two seasons (summer/fall and winter/spring) in order to account for seasonal variation in vitamin D status. Ca (2000 mg/d) and vitamin D (1000 IU/d) will be supplied as either capsules or a fortified food product daily throughout training. This study will provide novel data for the military, medical and scientific communities regarding the relationship between Ca and vitamin D supplementation and biomarkers of immune function, and the requirements for calcium and vitamin D to support bone health during IMT.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Marine Corps recruit at least 17 years of age.

Exclusion Criteria:

* Pregnant or breastfeeding
* History of kidney stones or kidney disease
* History of endocrine disorders
* Allergies to any component of the food product bar

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Serum Bone Health Biomarkers (Composite) | Measures will be taken at the beginning and end of Initial Military Training (IMT) which is approximately 12 weeks
  Effect of calcium/vitamin D on the following serum biomarkers:
  25(OH)D (ng/ml), parathyroid hormone (PTH) (pg/ml), C-telopeptide cross-links of type 1 collagen (CTX) (ng/ml), tartrate-resistant acid phosphatase (TRAP) (U/L), bone alkaline phosphatase (BAP) (ug/L), procollagen I N-terminal peptide (P1NP) (ug/L)

SECONDARY OUTCOMES:
Bone Strength Indices (Composite) | Measures will be taken at the beginning and end of Initial Military Training (IMT) which is approximately 12 weeks
  Effect of calcium/vitamin D on the following indices of bone strength as assessed by peripheral quantitative computed tomography (pQCT):
  volumetric bone mineral density (vBMD) (mg/cm3), bone strength index (BSI) (mg/mm4), cortical bone mineral content (Crt BMC) (mg/mm), cortical volumetric bone mineral density (Crt vBMD) (mg/cm3), strength strain index (SSI) (no units)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Gaffney-Stomberg, Ph.D., R.D., Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- Marine Corps Recruit Depot Parris Island, Parris Island, South Carolina, United States

REFERENCES:
- [Derived] Nakayama AT, Lutz LJ, Hruby A, Karl JP, McClung JP, Gaffney-Stomberg E. A dietary pattern rich in calcium, potassium, and protein is associated with tibia bone mineral content and strength in young adults entering initial military training. Am J Clin Nutr. 2019 Jan 1;109(1):186-196. doi: 10.1093/ajcn/nqy199. PMID 30615068